CLINICAL TRIAL: NCT03069482
Title: Feasibility Trial of a Tailored Smoking Cessation App for People With Serious Mental Illness
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00075165; 4R00DA037276-03 (NIH)
Record Dates: First submitted 2017-02-22; First posted 2017-03-03 (Actual); Results first posted 2020-03-23 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-10

CONDITIONS: Nicotine Addiction; Serious Mental Illness
Keywords: Smoking; mHealth; Serious Mental Illness; Acceptance and Commitment Therapy; US DHHS Clinical Practice Guidelines
MeSH Terms: conditions — Tobacco Use Disorder; Smoking | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Intervention Model Description: Subjects will be assigned to one of two smoking cessation apps for the duration of the study: Learn to Quit or NCI QuitGuide. One app was designed to address the needs of people with serious mental illness (Learn to Quit) and the other was designed for the general population (NCI QuitGuide).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Learn to Quit (Experimental): A smartphone app developed by the research team designed for people with serious mental illness, that provides Acceptance and Commitment Therapy skills to address (a) smoking cessation and (b) mental health symptoms.
  Interventions: Device: Learn to Quit App; Drug: Nicotine patch; Drug: Nicotine lozenge; Behavioral: Technical Coaching
- NCI QuitGuide (Active Comparator): A smartphone app developed by the National Cancer Institute which uses smoking cessation recommendations contained in the US DHHS Clinical Practice Guidelines.
  Interventions: Drug: Nicotine patch; Drug: Nicotine lozenge; Behavioral: Technical Coaching; Device: NCI QuitGuide App

INTERVENTIONS:
Device: Learn to Quit App — A smartphone app designed for individuals with serious mental illness. The main intervention components of the app are skills based on an intervention called Acceptance and Commitment Therapy that will (a) teach smoking cessation skills and (b) help cope with mental health symptoms. The app incorporates gaming features to keep users engaged, and a tracking component to record smoking habits and moods.
  Arms: Learn to Quit
Drug: Nicotine patch — Participants enrolled in the study will be given an 8-week course of Nicotine patches. The 8-week course of trans-dermal nicotine patches starting at 21mg/24h for 4 weeks, then transitioning to 14mg/24h for 2 weeks, and finally to 7mg/24h for the last 2 weeks. This dosing will follow recommendations contained in the US DHHS Clinical Practice Guidelines.
Drug: Nicotine lozenge — Each participant will be given a 1-week course of 4mg Nicotine lozenges to be taken orally as nicotine cravings arise (about 10 lozenges per day). They will be directed to use them for the week following their quit date, using no more than once every 1-2 hours. This dosing will follow recommendations contained in the US DHHS Clinical Practice Guidelines.
Behavioral: Technical Coaching — Coaching to assist the user on the use of each assigned smartphone app. This coaching will be delivered by research staff following a coaching procedure. These in-person coaching meetings will be brief (~15 minutes), done on a weekly basis for 4 weeks, and will have a focus on providing technical assistance.
Device: NCI QuitGuide App — A smartphone app developed by the National Cancer Institute which uses recommendations contained in the US DHHS Clinical Practice Guidelines and smokefree.gov. NCI QuitGuide has the following intervention components: (a) psycho-education about the impact of smoking in health, (b) tracking of smoking habits, and (c) Tips for quitting (e.g., distraction strategies).
  Arms: NCI QuitGuide

SUMMARY:
Quitting smoking has important health benefits for people with serious mental illness, more than half of whom are smokers. Smoking reductions in this population, in turn, could contribute to saving billions of dollars in healthcare expenditures.

Finding ways to deliver more effective and wider reaching smoking cessation interventions to individuals with serious mental illness is a pressing priority. Smartphone apps are a wide reaching technology that could provide a viable platform to deliver smoking cessation interventions for individuals with serious mental illness.

However, do smoking cessation apps need to be tailored for people with serious mental illness to ensure their success? Or can providers simply use standard and freely available smoking cessation mobile health treatments designed for the general population? Furthermore, is it feasible to conduct mHealth trials in this population?

Therefore, this trial will test whether (1) a tailored smoking cessation app for people with serious mental illness results in higher levels of engagement with smoking cessation content as compared to an app designed for the general population and (2) smoking cessation mHealth trials can be feasibly conducted in this population.

DETAILED DESCRIPTION:
Smoking tobacco shortens the lifespan of adults with serious mental illness by 25 years and contributes to $317 billion expenditures in healthcare, indirect loss of earnings and disability benefits. Determining whether it is possible to deliver more effective and wider reaching smoking cessation interventions to individuals with serious mental illness is a high priority. Smartphone apps are a wide reaching technology that could provide individuals with serious mental illness the necessary skills for quitting.

This feasibility trial will test whether a tailored smoking cessation app for people with serious mental illness, Learn to Quit, results in higher levels of engagement with smoking cessation content as compared to an app designed for the general population, NCI QuitGuide. The trial will also demonstrate whether it is possible to (a) feasibly recruit and retain individuals with serious mental illness in an mHealth clinical trial, and (b) successfully gather smoking cessation outcomes. Ninety individuals with serious mental illness will be randomly assigned to one of two conditions. In the experimental condition, participants will use the Learn to Quit app. In the comparator condition, participants will use the NCI QuitGuide app. Participants in both conditions will receive Nicotine Replacement Therapy (standard dosing of nicotine patch + 1-week course of 4mg nicotine lozenges) and technical coaching. Study duration will be 4 months, with four follow-up appointments at 1-month, 2-month, 3-month, and 4-months.

ELIGIBILITY:
Inclusion Criteria:

* ICD-10 diagnosis of schizophrenia, schizoaffective, bipolar or recurring depressive disorder
* Smoking ≥ 5 cigarettes per day over the past 30 days
* Desire to quit smoking in the next 30 days
* Willing and medically eligible to use Nicotine Replacement Therapy
* Fluent in spoken and written English
* Working email, mailing address, or alternative contact person
* Taking psychiatric medications as prescribed by their provider
* Stable housing

Exclusion Criteria:

* Problematic alcohol or illicit drug use in the last 30 days
* Acute psychotic episode, unsafe to participate in the study, or psychiatrically unstable
* Pregnant, breastfeeding, or having the intention to become pregnant in the next 4 months
* Hearing, comprehension, or visual limitations that preclude study participation
* Currently receiving any pharmacological and/or behavioral intervention or counseling for smoking cessation
* Using non-cigarette forms of tobacco as the primary source of nicotine (e.g. e-cigarettes, chew)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2019-01-17 (Actual); Study Completion 2019-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Vilardaga, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Browne J, Halverson TF, Vilardaga R. Engagement with a digital therapeutic for smoking cessation designed for persons with psychiatric illness fully mediates smoking outcomes in a pilot randomized controlled trial. Transl Behav Med. 2021 Sep 15;11(9):1717-1725. doi: 10.1093/tbm/ibab100. PMID 34347865

RESULTS

PARTICIPANT FLOW:
Groups:
- Learn to Quit: A smartphone app developed by the research team designed for people with serious mental illness, that provides Acceptance and Commitment Therapy skills to address (a) smoking cessation and (b) mental health symptoms. This app intervention is combined with an 8-week course of nicotine replacement therapy (NRT) patches and a 2-week course of NRT lozenges. Participants also receive technical smartphone coaching for the first 4 weeks of the study.
- NCI QuitGuide: A smartphone app developed by the National Cancer Institute which uses smoking cessation recommendations contained in the US DHHS Clinical Practice Guidelines. The app intervention is combined with an 8-week course of nicotine replacement therapy (NRT) patches and a 2-week course of NRT lozenges. Participants also receive technical smartphone coaching for the first 4 weeks of the study.
Period: Overall Study
Arm/Group | Learn to Quit | NCI QuitGuide
Started | 34 | 29
Completed | 33 | 28
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: One participant (Learn to Quit arm) was withdrawn by physician and therefore was not included in these analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Learn to Quit | NCI QuitGuide | Total
Number analyzed (Participants) | 33 | 29 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 29 | 60
  >=65 years | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (11.2) | 45.6 (10.9) | 47.1 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 16 | 37
  Male | 12 | 13 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 33 | 28 | 61
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 11 | 25
  White | 16 | 16 | 32
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 33 | 29 | 62
CPD at Baseline [Mean (Standard Deviation); unit: cigarettes per day] — Number of average cigarettes smoked per day at baseline.
  cigarettes per day | 21 (15.5) | 14 (6.4) | 17.9 (12.6)
MDD Diagnosis [Count of Participants; unit: Participants] — Percentage of participant enrolled who had a diagnosis of recurrent major depressive disorder.
  Participants | 8 | 9 | 17
Bipolar Diagnosis [Count of Participants; unit: Participants] — Percentage of participants enrolled who had diagnosis of bipolar I or II disorder.
  Participants | 15 | 15 | 30
Schizophrenia Spectrum Diagnosis [Count of Participants; unit: Participants] — Percentage of participants enrolled who had a diagnosis of schizophrenia or schizoaffective disorder.
  Participants | 10 | 5 | 15
Education Levels [Count of Participants; unit: Participants] — The highest level of education by participants completed across groups.
  Participants
    Secondary School or Less | 11 | 10 | 21
    Some College | 9 | 8 | 17
    Associate's Degree | 4 | 5 | 9
    Bachelor's Degree or Higher | 9 | 6 | 15
Disability Status [Count of Participants; unit: Participants] — Number of participants who self-reported to be on employment disability across groups.
  Participants | 19 | 9 | 28
Years of Smoking [Mean (Standard Deviation); unit: years] — Self-reported years of everyday smoking across groups
  years | 25.6 (12.9) | 26.8 (11.3) | 26.2 (12.1)
Nicotine Dependence [Mean (Standard Deviation); unit: units on a scale] — Nicotine dependence across groups as determined by the Fagerstrom Test for Nicotine Dependence. Scores range from 0 to 11 with higher scores indicating higher nicotine dependence.
  units on a scale | 5.2 (2.6) | 4.7 (2.3) | 5.0 (2.5)
Cognitive Functioning [Mean (Full Range); unit: units on a scale] — Cognitive functioning as assessed by the Brief Assessment of Cognition. Means are represented as Z-scores (lower scores = lower cognitive functioning, higher scores = higher cognitive functioning).
  units on a scale | -1 [-3.73 to 1.66] | -0.9 [-5.19 to 1.20] | -0.95 [-5.19 to 1.66]
Household Income [Count of Participants; unit: Participants] — Self-reported combined yearly income for all members living in the participants' households, across groups.
  Participants
    <$35,000 | 24 | 18 | 42
    $35-50,0000 | 4 | 2 | 6
    $50-75,000 | 0 | 4 | 4
    $75-100,000 | 1 | 1 | 2
    >$100,000 | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Days of App Use
Description: Frequency of app openings in each group
Time Frame: Daily throughout study duration, 4 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 33 | 29
days | 34.1 (27.7) | 32 (24.5)
Statistical Analysis 1: Comparison: Learn to Quit vs NCI QuitGuide; Test type: Superiority; p = 0.754, ANOVA; Slope = 1.063, Standard Deviation 3.377

2. Primary Outcome: Duration of App Use
Description: Mean duration of app use in each group over the course of study participation (4 months)
Time Frame: Daily throughout study duration, 4 months
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 33 | 29
hours | 4.24 (4.29) | 2.14 (1.72)
Statistical Analysis 1: Comparison: Learn to Quit vs NCI QuitGuide; Test type: Superiority; p = 0.044, Mixed Models Analysis; Zero inflated negative binomial mixed methods regression; Risk Ratio (RR) = 2.103, 095% CI 2-sided [1.2 to 2.6], Standard Deviation 0.369

3. Primary Outcome: Feasibility as Measured by Study Accrual Relative to Recruitment Goal
Description: Percent of subjects consented into study relative to study recruitment goal (N=90).92 subjects signed consent prior to eligibility determination and randomization.
Time Frame: Approximately 15 months
Population: The number of participants analyzed in this sample is larger than the number of participants who were ultimately randomized to the study as reflected in the participant flow section. This sample includes all participants who were consented into the study regardless of their final eligibility status prior to randomization.
Measure: Number; unit: percentage of target accrual
Groups:
- All Consented Participants: All participants consented to the study prior to eligibility determination.
Arm/Group | All Consented Participants
Number analyzed (Participants) | 92
percentage of target accrual | 102
Statistical Analysis 1: Comparison: All Consented Participants; Test type: Other; Percent accrual relative to target N = 102; The goal of this outcome was to determine whether the trial could reach its enrollment target (90 participants)

4. Primary Outcome: Feasibility as Measured by Study Attrition
Description: Number and percentage of subjects who complete 4-month follow up assessment
Time Frame: 4-months
Measure: Count of Participants; unit: Participants
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 33 | 29
Participants | 33 | 28
Statistical Analysis 1: Comparison: Learn to Quit vs NCI QuitGuide; Test type: Other; Percent retention relative to target = 98.3; We calculated the percent of retained participants relative to the retention target (N = 62)

5. Primary Outcome: Recruitment Yield Effort
Description: Percent of subjects responding to ads and clinician referrals
Time Frame: Approximately 15 months
Measure: Count of Participants; unit: Participants
Groups:
- Total Patients in Database: The total amount of patients who could have potentially contacted us or that we could have approached to participate in the study.
Arm/Group | Total Patients in Database
Number analyzed (Participants) | 499
Participants | 290
Statistical Analysis 1: Comparison: Total Patients in Database; Test type: Other; Percent of respondents = 58

6. Primary Outcome: Feasibility of Measurement Strategy
Description: Percent completion of assessment measures. Assessment measures include surveys, questionnaires, and cognitive tasks.
Time Frame: Approximately 19 months
Population: Number of total possible assessment measures that could have been completed in each group.
Measure: Count of Units; unit: assessments
Units Other Than Participants: assessments
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 33 | 29
Number analyzed (assessments) | 1617 | 1421
assessments | 1353 | 1284

7. Primary Outcome: Usability of App Design as Measured by the System Usability Scale (SUS)
Description: 10-item scale giving a global assessment of systems usability using a 5-point Likert Scale with a composite score ranging from 0-100. Higher scores indicate higher usability rating.
Time Frame: 1-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 33 | 29
score on a scale | 87.3 (13.6) | 79.4 (15)
Statistical Analysis 1: Comparison: Learn to Quit vs NCI QuitGuide; Test type: Superiority; p = 0.046, Yuen's trimmed mean t-test; Trimmed mean difference = 8.29574, 95% CI 2-sided [0.138 to 16.453], Standard Error of Mean 2.11

8. Primary Outcome: Usability of App Design as Measured by the System Usability Scale (SUS)
Description: as for outcome 7
Time Frame: 2-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 33 | 29
score on a scale | 84.4 (13.5) | 75.6 (19.6)
Statistical Analysis 1: Comparison: Learn to Quit vs NCI QuitGuide; Test type: Superiority; p = 0.109, Yuen's trimmed means t-test; Trimmed mean difference = 7.79514, 95% CI 2-sided [-1.867 to 17.457], Standard Error of Mean 2.16

9. Primary Outcome: Usability of App Design as Measured by the System Usability Scale (SUS)
Description: as for outcome 7
Time Frame: 3-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 33 | 29
score on a scale | 83.2 (14.1) | 80.8 (15.6)
Statistical Analysis 1: Comparison: Learn to Quit vs NCI QuitGuide; Test type: Superiority; p = 0.50537, Yuen's trimmed means t-test; Trimmed mean difference = 2.22222, 95% CI 2-sided [-4.492 to 8.943], Standard Error of Mean 1.75

10. Primary Outcome: Usability of App Design as Measured by the System Usability Scale (SUS)
Description: as for outcome 7
Time Frame: 4-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 33 | 29
score on a scale | 85.2 (13.9) | 78.7 (19.3)
Statistical Analysis 1: Comparison: Learn to Quit vs NCI QuitGuide; Test type: Superiority; p = 0.27411, Yuen's trimmed means t-test; Trimmed mean difference = 5.83333, 95% CI 2-sided [-4.88 to 16.54], Standard Error of Mean 2.30

11. Secondary Outcome: Biochemically Confirmed 7-day Point Prevalence Abstinence
Description: Percent of subjects in each group reporting biochemically confirmed 7-day point prevalence abstinence. Abstinence is determined by a self-report of not smoking for 7 days prior to the specified timepoint AND by a result of ≤ 5 ppm in carbon monoxide breath testing. If the participant does not meet both criteria, they are not considered abstinent.
Time Frame: 1 month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 33 | 29
Participants | 3 | 5

12. Secondary Outcome: Biochemically Confirmed 7-day Point Prevalence Abstinence
Description: as for outcome 11
Time Frame: 2 month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 33 | 29
Participants | 6 | 0

13. Secondary Outcome: Biochemically Confirmed 7-day Point Prevalence Abstinence
Description: as for outcome 11
Time Frame: 3 month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 33 | 29
Participants | 3 | 2

14. Secondary Outcome: Biochemically Confirmed 7-day Point Prevalence Abstinence
Description: as for outcome 11
Time Frame: 4 month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 33 | 29
Participants | 4 | 1

15. Secondary Outcome: Biochemically Confirmed Prolonged Abstinence Rates
Description: Total number of participants in each group reporting prolonged abstinence at the specified time point. Abstinence is determined by a self-report of not relapsing after their quit date (i.e., not smoking for 7 consecutive days, or not smoking at least once each week for 2 consecutive weeks) following a 2-week grace period, AND by a result of ≤ 6 ppm in carbon monoxide breath testing. If the participant does not meet both criteria, they are not considered abstinent
Time Frame: 1 month follow up
Population: A survey branching logic error led to incomplete data collection for this measure. Therefore, we could not collect data from all participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 11 | 15
Participants | 4 | 3

16. Secondary Outcome: Biochemically Confirmed Prolonged Abstinence Rates
Description: as for outcome 15
Time Frame: 2 month follow up
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 5 | 6
Participants | 0 | 0

17. Secondary Outcome: Biochemically Confirmed Prolonged Abstinence Rates
Description: as for outcome 15
Time Frame: 3 month follow up
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 6 | 3
Participants | 0 | 0

18. Secondary Outcome: Biochemically Confirmed Prolonged Abstinence Rates
Description: as for outcome 15
Time Frame: 4 month follow up
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 3 | 4
Participants | 0 | 0

19. Secondary Outcome: 30-day Point Prevalence Abstinence Rates
Description: Participants who self-reported not smoking for 30 days prior to the specified timepoint.
Time Frame: 1 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 33 | 29
Participants | 0 | 1

20. Secondary Outcome: 30-day Point Prevalence Abstinence Rates
Description: Participants who self-reported not smoking for 30 days prior to the specified timepoint.
Time Frame: 2 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 33 | 29
Participants | 3 | 2

21. Secondary Outcome: 30-day Prevalence Abstinence Rates
Description: Participants who self-reported not smoking for 30 days prior to the specified timepoint.
Time Frame: 3 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 33 | 29
Participants | 1 | 3

22. Secondary Outcome: 30-day Point Prevalence Abstinence Rates
Description: Participants who self-reported not smoking for 30 days prior to the specified timepoint.
Time Frame: 4 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 33 | 29
Participants | 4 | 3

23. Secondary Outcome: 7-day Point Prevalence Abstinence
Description: Participants who self-reported not smoking for 7 days prior to the specified timepoint.
Time Frame: 1 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 33 | 29
Participants | 4 | 7

24. Secondary Outcome: 7-day Point Prevalence Abstinence
Description: Participants who self-reported not smoking for 7 days prior to the specified timepoint.
Time Frame: 2 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 33 | 29
Participants | 6 | 2

25. Secondary Outcome: 7-day Point Prevalence Abstinence
Description: Participants who self-reported not smoking for 7 days prior to the specified timepoint.
Time Frame: 3 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 33 | 29
Participants | 5 | 4

26. Secondary Outcome: 7-day Point Prevalence Abstinence
Description: Participants who self-reported not smoking for 7 days prior to the specified timepoint.
Time Frame: 4 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 33 | 29
Participants | 4 | 3

27. Secondary Outcome: 24-hour Point Prevalence Abstinence
Description: Participants who self-reported not smoking for 24 hours prior to the specified timepoint.
Time Frame: 1 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 33 | 29
Participants | 8 | 10

28. Secondary Outcome: 24-hour Point Prevalence Abstinence
Description: Participants who self-reported not smoking for 24 hours prior to the specified timepoint.
Time Frame: 2 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 33 | 29
Participants | 8 | 7

29. Secondary Outcome: 24-hour Point Prevalence Abstinence
Description: Participants who self-reported not smoking for 24 hours prior to the specified timepoint.
Time Frame: 3 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 33 | 29
Participants | 6 | 6

30. Secondary Outcome: 24-hour Point Prevalence Abstinence
Description: Participants who self-reported not smoking for 24 hours prior to the specified timepoint.
Time Frame: 4 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 33 | 29
Participants | 7 | 7

31. Secondary Outcome: Average Number of Quit Attempts Per Arm
Description: Average number of quit attempts per group defined as self-reported no smoking at all for 24 hours at the specified time point.
Time Frame: 1 month follow up
Measure: Mean (Standard Deviation); unit: quit attempts
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 33 | 29
quit attempts | 1.16 (1.19) | 3.04 (2.29)

32. Secondary Outcome: Average Number of Quit Attempts Per Arm
Description: as for outcome 31
Time Frame: 2 month follow up
Measure: Mean (Standard Deviation); unit: quit attempts
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 33 | 29
quit attempts | 1.44 (1.34) | 2.55 (1.82)

33. Secondary Outcome: Average Number of Quit Attempts Per Arm
Description: as for outcome 31
Time Frame: 3 month follow up
Measure: Mean (Standard Deviation); unit: quit attempts
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 33 | 29
quit attempts | 1.83 (2.17) | 3.30 (3.61)

34. Secondary Outcome: Average Number of Quit Attempts Per Arm
Description: as for outcome 31
Time Frame: 4 month follow up
Measure: Mean (Standard Deviation); unit: quit attempts
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 33 | 29
quit attempts | 1.61 (1.85) | 1.96 (1.90)

35. Secondary Outcome: Change in Nicotine Dependence as Measured by the Fagerstrom Test of Nicotine Dependence
Description: The Fagerstrom Test of Nicotine Dependence ranges from 0 to 10 with the lower score indicating "no dependence" and the highest score indicating "very dependent"
Time Frame: Baseline to 1, 2, 3 and 4 month follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 33 | 29
units on a scale
  Week 4 | 0.81 (2.17) | 1.88 (2.90)
  Week 8 | 1 (1.97) | 1.47 (2.67)
  Week 12 | 1.29 (2.03) | 1.74 (2.40)
  Week 16 | 1.16 (2.03) | 1.35 (2.48)

36. Secondary Outcome: Change in Average Number of Cigarettes Smoked Per Day
Description: Change in average number of self-reported cigarettes smoked per day per arm from baseline to the specified time point.
Time Frame: Baseline to 1, 2, 3 and 4 month follow up
Measure: Mean (Standard Deviation); unit: cigarettes per day
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 33 | 29
cigarettes per day
  Week 4 | 10.0 (9.9) | 5.2 (10.8)
  Week 8 | 11.3 (12.0) | 7.5 (7.6)
  Week 12 | 11.5 (12.3) | 6.0 (7.6)
  Week 16 | 12.3 (11.5) | 5.9 (5.9)

37. Secondary Outcome: Nicotine Replacement Patch Utilization
Description: Days of patch use over the last 30 days.
Time Frame: 1 month follow up
Measure: Mean (Standard Deviation); unit: days of patch use
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 33 | 29
days of patch use | 10.3 (10.4) | 13.9 (11.6)

38. Secondary Outcome: Nicotine Replacement Patch Utilization
Description: Days of patch use over the last 30 days.
Time Frame: 2 month follow up
Measure: Mean (Standard Deviation); unit: days of patch use
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 33 | 29
days of patch use | 11 (11.2) | 14.9 (12.8)

39. Secondary Outcome: Nicotine Replacement Patch Utilization
Description: Days of patch use over the last 30 days.
Time Frame: 3 month follow up
Measure: Mean (Standard Deviation); unit: days of patch use
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 33 | 29
days of patch use | 8.4 (10.7) | 7.4 (9.5)

40. Secondary Outcome: Nicotine Replacement Patch Utilization
Description: Days of patch use over the last 30 days.
Time Frame: 4 month follow up
Measure: Mean (Standard Deviation); unit: days of patch use
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 33 | 29
days of patch use | 3.4 (6.2) | 5.3 (8.6)

41. Secondary Outcome: Nicotine Replacement Lozenge Utilization
Description: Days of lozenge use over the last 30 days.
Time Frame: 1 month follow up
Measure: Mean (Standard Deviation); unit: days of lozenge use
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 33 | 29
days of lozenge use | 7.8 (9.7) | 10 (10)

42. Secondary Outcome: Nicotine Replacement Lozenge Utilization
Description: Days of lozenge use over the last 30 days.
Time Frame: 2 month follow up
Measure: Mean (Standard Deviation); unit: days of lozenge use
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 33 | 29
days of lozenge use | 5.1 (9.3) | 7 (10.4)

43. Secondary Outcome: Nicotine Replacement Lozenge Utilization
Description: Days of lozenge use over the last 30 days.
Time Frame: 3 month follow up
Measure: Mean (Standard Deviation); unit: days of lozenge use
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 33 | 29
days of lozenge use | 4.4 (8) | 4.1 (7.2)

44. Secondary Outcome: Nicotine Replacement Lozenge Utilization
Description: Days of lozenge use over the last 30 days.
Time Frame: 4 month follow up
Measure: Mean (Standard Deviation); unit: days of lozenge use
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 33 | 29
days of lozenge use | 2.3 (6.3) | 1.3 (3.1)

45. Secondary Outcome: Affect Ratings - Learn to Quit
Description: Average mood rating as self-reported through the Learn to Quit app. Ratings range from 1-10 with lower scores indicating poorer mood ratings.
Time Frame: Daily throughout study duration, 4 months
Population: Participants in the Learn to Quit group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Learn to Quit
Number analyzed (Participants) | 33
score on a scale | 5.4666165 (2.155668)

46. Secondary Outcome: Affect Ratings - QuitGuide
Description: Percent of reported positive, negative, and mixed affect. Negative affect was coded as '1' when the following types of mood were reported using the mood tracking feature within the app: frustrated, stressed, nervous, anxious, angry, sad. Positive affect was coded as '1' when the following types of mood were reported using the mood tracking feature within the app: happy, relaxed, excited. Mixed affect was coded as '1' when there were instances where participants reported both positive and negative affect at different times of the day.
Time Frame: Daily throughout study, 4 months
Population: Participants in the QuitGuide group.
Measure: Number; unit: Percent of counts
Groups:
- QuitGuide: A smartphone app developed by the National Cancer Institute which uses smoking cessation recommendations contained in the US DHHS Clinical Practice Guidelines. The app intervention is combined with an 8-week course of nicotine replacement therapy (NRT) patches and a 2-week course of NRT lozenges. Participants also receive technical smartphone coaching for the first 4 weeks of the study.
Arm/Group | QuitGuide
Number analyzed (Participants) | 29
Percent of counts
  Positive Affect | 52.26
  Negative Affect | 43.90
  Mixed Affect | 3.83

47. Secondary Outcome: Smoking Cravings
Description: Average daily smoking cravings as self-reported through each smartphone app. Cravings range from a score of 1 to 10 with higher scores indicating higher cravings to smoke.
Time Frame: Daily throughout study duration, 4 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 33 | 29
units on a scale | 6.13 (2.25) | 4.55 (2.98)

48. Secondary Outcome: Psychotic Symptoms
Description: Psychotic symptoms (positive and negative symptoms) at the specified time point as measured by the Positive and Negative Symptoms Scale. Scores range from 7 to 49 with higher scores indicating more psychopathology.
Time Frame: 1 month follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 33 | 29
score on a scale
  Positive symptoms | 11.74 (3.43) | 11.85 (3.52)
  Negative symptoms | 11.61 (4.38) | 10.81 (4.33)

49. Secondary Outcome: Psychotic Symptoms
Description: as for outcome 48
Time Frame: 2 month follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 33 | 29
score on a scale
  Positive symptoms | 11.55 (3.49) | 10.79 (3.79)
  Negative symptoms | 12.45 (4.42) | 11.38 (5.38)

50. Secondary Outcome: Psychotic Symptoms
Description: as for outcome 48
Time Frame: 3 month follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 33 | 29
score on a scale
  Positive symptoms | 11.10 (4.21) | 12.32 (5.00)
  Negative symptoms | 12.57 (5.82) | 12.25 (5.08)

51. Secondary Outcome: Psychotic Symptoms
Description: as for outcome 48
Time Frame: 4 month follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 33 | 29
score on a scale
  Positive symptoms | 11.63 (4.53) | 11.55 (3.86)
  Negative symptoms | 12.16 (4.25) | 12.23 (5.23)

52. Secondary Outcome: General Psychiatric Symptoms
Description: General psychiatric symptoms at the specified time point as measured by the Global Severity Index of the Brief Symptom Inventory. Scores range from 0 to 4 with higher scores indicating more psychiatric symptoms.
Time Frame: 1 month follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 33 | 29
score on a scale | 0.92 (0.59) | 0.84 (0.65)

53. Secondary Outcome: General Psychiatric Symptoms
Description: as for outcome 52
Time Frame: 2 month follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 33 | 29
score on a scale | 0.87 (0.64) | 0.68 (0.58)

54. Secondary Outcome: General Psychiatric Symptoms
Description: as for outcome 52
Time Frame: 3 month follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 33 | 29
score on a scale | 0.80 (0.58) | 0.80 (0.60)

55. Secondary Outcome: General Psychiatric Symptoms
Description: as for outcome 52
Time Frame: 4 month follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Learn to Quit | NCI QuitGuide
Number analyzed (Participants) | 33 | 29
score on a scale | 0.94 (0.75) | 0.90 (0.64)

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Learn to Quit | NCI QuitGuide
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/29
Serious Adverse Events (participants affected / at risk) | 6/33 | 4/29
Other Adverse Events (participants affected / at risk) | 30/33 | 23/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Learn to Quit (N=33) | NCI QuitGuide (N=29)
Second degree burns (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Low blood pressure (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hospitalization from elevated blood sugar (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Heroin overdose (Social circumstances) | 0 (0) | 1 (1)
Withdrawal from methadone (Social circumstances) | 1 (1) | 0 (0)
Knee surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Hospitalized because of two broken arms (Surgical and medical procedures) | 1 (1) | 0 (0)
Hospitalization due to suicidal ideation (Psychiatric disorders) | 1 (2) | 0 (0)
Mini-stroke (TIA) (Nervous system disorders) | 1 (1) | 0 (0)
Asthma attack (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hernia repair surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Learn to Quit (N=33) | NCI QuitGuide (N=29)
Anxiety and stress (Psychiatric disorders) | 4 (4) | 4 (4) — Feeling anxious, stressed, or "on edge"
Dental procedures (Surgical and medical procedures) | 3 (3) | 1 (1)
Body aches and pains (Musculoskeletal and connective tissue disorders) | 6 (7) | 6 (6)
Changes in blood pressure (Vascular disorders) | 3 (4) | 1 (1)
Burning in mouth/throat/chest (Gastrointestinal disorders) | 3 (3) | 6 (6)
Broken/sprained body parts (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2)
Coughing (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 4 (5)
Cold/flu (Infections and infestations) | 6 (7) | 5 (8)
Acid reflux (Gastrointestinal disorders) | 0 (0) | 3 (3)
Allergies/asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (7) | 4 (4)
Itchy/irritated skin (Skin and subcutaneous tissue disorders) | 6 (7) | 6 (6)
Skin breakouts (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 3 (3) | 1 (1)
Nightmares/vivid dreams (Psychiatric disorders) | 1 (1) | 5 (5)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Sleep issues (Psychiatric disorders) | 2 (2) | 2 (2)
Frustration due to phone/app issues (Psychiatric disorders) | 1 (1) | 1 (1)
Infections (Infections and infestations) | 0 (0) | 2 (2)
Tumor removal (procedure) (Surgical and medical procedures) | 0 (0) | 1 (1)
Cyst/abcess removal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Accidents (Social circumstances) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lacerations (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Agoraphobia (Psychiatric disorders) | 0 (0) | 1 (1)
Aversion to NRT taste (Product Issues) | 1 (1) | 0 (0)
Headaches (General disorders) | 1 (1) | 2 (2)
Eye procedure (Surgical and medical procedures) | 1 (1) | 1 (1)
Reproductive problems (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cancer (General disorders) | 2 (2) | 0 (0)
Opioid withdrawal (Psychiatric disorders) | 1 (1) | 0 (0)
Vision problems (Eye disorders) | 2 (2) | 0 (0)
Congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Dry mouth while using lozenges (Product Issues) | 2 (2) | 0 (0)
Memory problems (Psychiatric disorders) | 0 (0) | 1 (1)
Changes in blood sugar levels (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Thyroid problems (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Sore throat (Infections and infestations) | 0 (0) | 1 (1)
Increased heart rate (Cardiac disorders) | 0 (0) | 1 (2)
Changes in mood (Psychiatric disorders) | 1 (1) | 2 (2)
Tooth pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
NRT adherence measure relied on self-report. Participant stratification did not successfully balance presence of mood vs. psychotic disorders in each group. 26% of outcomes measures collected via phone or web survey due to transportation barriers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-05): https://cdn.clinicaltrials.gov/large-docs/82/NCT03069482/Prot_SAP_000.pdf